CLINICAL TRIAL: NCT07052552
Title: Adding Ujjayi Pranayama to Osteopathic Manipulative Treatment on Pulmonary Functions and Functional Capacity in College Students With Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Mohamed Saied Zidan, Assistant professor doctor, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 2/6/2024-2025
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Osteopathic Manipulation; Ujjayi Pranayama; Upper Cross Syndrome
Keywords: Ujjayi pranayama; Osteopathic Manipulation; Upper cross syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): control group will perform osteopathic manipulative tratment only
  Interventions: Other: osteopathic manipulative tratment only
- Experimental group (Experimental): experimental group will perform ujjayi pranayama and osteopathic manipulative treatment
  Interventions: Other: ujjayi pranayama and osteopathic manipulative treatment

INTERVENTIONS:
Other: osteopathic manipulative tratment only — focuses on restoring proper muscle balance and joint mechanics through techniques that address the shortened, tight muscles and the lengthened, weak muscles characteristic of the syndrome
  Arms: Control group
Other: ujjayi pranayama and osteopathic manipulative treatment — Ujjayi pranayama, often called "ocean breath," can be a helpful practice for individuals with Upper Cross Syndrome (UCS) by promoting relaxation and improving breath control. While not a direct cure, it can alleviate some symptoms and improve overall posture and body awareness.
  Osteopathic manipulative treatment focuses on restoring proper muscle balance and joint mechanics through techniques that address the shortened, tight muscles and the lengthened, weak muscles characteristic of the syndrome
  Arms: Experimental group

SUMMARY:
With the advent of the Internet, mobile phones and other electronic devices have become an integral component in everyone's lives, especially students, whether it is to attend classes, make purchases, conduct transactions, or have social interactions . The continuous use of these electronic devices can easily result in abnormal postures . Upper crossed syndrome (UCS) is one of the most frequently cited complications with modern technological life, which is characterized by weakened middle and lower trapezius, scalenes, deep cervical flexors and serratus anterior at the same time as the rhomboids, as well as tightness in the upper trapezius, pectoralis minor and major and levator scapulae muscles . It mainly leads to muscle imbalances, which eventually manifest in both tonic and phasic muscles

ELIGIBILITY:
Inclusion Criteria:

* Full time college students of age 20-29 years.

  * Subjects who have upper cross syndrome according to REEDCO posture assessment.
  * Subjects who not receiving medical treatment for respiratory diseases .
  * Subjects who have clean family medical history

Exclusion Criteria:

* Subjects who engaged in additional exercise in two weeks, which was likely to affect the results of the research .

  * Individuals with a history of spine, shoulder fractures, surgery, or other disease.
  * Individuals with severe cardia-cerebrovascular disease.
  * Individuals who will have difficulty to follow-up testing).
  * Neurologic and psychiatric disorders (who can not understand the research project ).
  * Individuals with congenital deformities

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
FVC ( liters ) | Pre and post 8 weeks
  Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test. Forced expiratory volume and forced vital capacity are lung function tests , using portable spirometer ( SP 80B , China )
FEV1 ( liters ) | Pre and post 8 weeks
  Forced expiratory volume in 1 second that can reflect pulmonary function , using portable spirometer ( SP 80B,China)
FEV1/FVC ( % ) | pre and post 8 weeks
  The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. That can reflect pulmonary function , using portable spirometer ( SP 80B,China)
PEF ( liters / minute ) | pre and post 8 weeks
  Peak expiratory flow (PEF), a key indicator of lung function,using portable spirometer ( SP 80B,China)
Expiratory reserve volume ( ERV ) ( Liters ) | pre and post 8 weeks
  is the maximum amount of air that can be forcefully exhaled after a normal, tidal exhalation
maximum voluntary ventilation (MVV) ( liters/minute ) | Pre and post 8 weeks
  is a pulmonary function test that measures the maximum amount of air a person can breathe in and out of their lungs in one minute
The inspiratory reserve volume (IRV) ( Liters ) | Pre and post 8 weeks
  It represents the maximum amount of air that can be inhaled after a normal inhalation

SECONDARY OUTCOMES:
6MWDT ( meters ) | Pre and post 8 weeks
  focus on endurance and distance covered during a timed walk, rather than assessing the specific muscle imbalances and postural deviations characteristic of Upper Cross Syndrome
Timed up and go test ( seconds ) | Pre and post 8 weeks
  A simple, quick, and widely used clinical performance-based measure of functional mobility and fall risk. It assesses how long it takes for a person to rise from a chair, walk three meters, turn, walk back, and sit down again.
Berg Balance Scale (BBS) to test dynamic balance | Pre and post 8 weeks
  A widely used assessment tool in physical therapy to evaluate a patient's functional balance and fall risk. It consists of 14 tasks, scored on a 5-point scale from 0 to 4, with a total possible score of 56. A lower score indicates a higher risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Saied Zidan, Cairo, Egypt